CLINICAL TRIAL: NCT02079285
Title: Prospective Evaluation of the Yield and Diagnostic Accuracy of Endoscopic Ultrasound-guided Fine Needle Aspiration and Biopsy in the Absence of Rapid Onsite Evaluation
Brief Title: Prospective Evaluation of Diagnostic Accuracy of Endoscopic Ultrasound-guided Fine Needle Aspiration and Biopsy (EUS-FNAB) in the Absence of Rapid Onsite Evaluation
Acronym: FNASROSE
Status: Completed | Type: Observational
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Hong Joo Kim, MD, Kangbuk Samsung Hospital
Other Study IDs: FNASROSE
Record Dates: First submitted 2014-03-02; First posted 2014-03-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EUS-FNA: Any patients who will undergo EUS-FNA for pancreas lesion during the study period
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA

SUMMARY:
<Background/aims> Rapid onsite evaluation (ROSE) of endoscopic ultrasound-guided fine needle aspiration and biopsy (EUS-FNAB) specimens by attending cytopathologists has been demonstrated to improve diagnostic yields of EUS-FNAB. The practice of ROSE, however, varies across EUS programs in Unites States, Europe and other areas of world. The investigators have a plan to perform prospective evaluation of the yield of EUS-FNAB in the absence of ROSE, in which the adequacy of specimens will be assessed by a single endosonographer.

<Methods> All EUS-FNAB procedures will be performed by an experienced endosonographer and the adequacy of specimens obtained during EUS-FNAB will be also assessed by a same endosonographer. A specimen will be considered adequate if there is an adequate number of representative cells from the lesion. Samples considered to be adequate will be then interpreted as malignancy, highly atypical suggestive of malignancy, atypical favor reactive change, or negative for malignancy. Performance characteristics of EUS-FNAB including sensitivity, specificity, and accuracy will be determined by comparing EUS-FNAB results with the final diagnoses of the lesions, based upon the surgical pathology or clinical follow-up of more than 6 months with repeat imagings.

ELIGIBILITY:
Inclusion Criteria:

* Any patients who will undergo EUS-FNA for the diagnostic evaluation of pancreas lesion

Exclusion Criteria:

* Patients who refuse to undergo EUS-FNA

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients who will undergo EUS-FNA for the diagnostic evaluation of pancreas lesion
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy of EUS-FNA without ROSE | 7 days
  Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of EUS-FNA without ROSE

SECONDARY OUTCOMES:
Adequacy of obtained cytologic specimens | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sungkyunkwan University Kangbuk Samsung Hospital, Seoul, South Korea